CLINICAL TRIAL: NCT06997120
Title: Effectiveness and Implementation of a Meditation App Addressing Substance Use, Sexual Health, and Emotion Regulation Among Legal-Involved Youth
Brief Title: Testing the Effectiveness and Implementation of a Meditation App for Youth in the Legal System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Ashley D Kendall, Principal Investigator, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-0066; R01DA061795 (NIH)
Record Dates: First submitted 2025-05-20; First posted 2025-05-30 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Behavioral Health
Keywords: Juvenile legal system; Meditation; Mindfulness; Smartphone; Mobile health (mHealth); Ecological momentary assessment (EMA); Substance use; Mental health
MeSH Terms: conditions — Substance-Related Disorders; Psychological Well-Being | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants will be individually randomized at a 1:1 ratio to 1 of 2 smartphone app conditions: (1) Bodhi AIM (Action In Mindfulness), a 30-day meditation app, or (2) HIB (Health In Balance), a health promotion control app matched to Bodhi AIM for time and structure.
Who Masked: Outcomes Assessor
Masking Description: Both participants and outcome assessors will be blind to condition through completion of the baseline assessment including the first week-long EMA burst. Condition will become apparent to both participants and assessors at the time of app download, but will not be revealed to assessors at either of the follow-up time points until after the quantitative measures are complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bodhi AIM (Experimental): Participants randomized to the intervention arm will receive the Bodhi AIM meditation app.
  Interventions: Behavioral: Bodhi AIM (intervention group)
- HIB (Active Comparator): Participants randomized to the active control arm will receive the HIB health promotion app.
  Interventions: Behavioral: HIB (control group)

INTERVENTIONS:
Behavioral: Bodhi AIM (intervention group) — AIM (Action In Mindfulness) is a smartphone app that teaches users to establish a daily meditation practice via a 30-day "path," with each day consisting of a brief audio- or video-guided file. In addition to the 30 daily path files, users have access to a menu of "to go" audio-guided meditation practices that they may access any time to prepare for particular situations.
  Arms: Bodhi AIM
Behavioral: HIB (control group) — HIB (Health In Balance) is a smartphone app that is matched to AIM for time and structure, but includes health promotion content (e.g., educational information on substance use) in place of the meditation content featured in AIM. Like AIM, HIB includes a 30-day "path" of audio and video files, along with a menu of "to go" audio files that users may access any time to review key intervention concepts.
  Arms: HIB

SUMMARY:
The goals of this hybrid type 2 randomized controlled trial (RCT) are to evaluate the effectiveness and individual-level implementation of a 1-month app-based meditation program with youth on probation in Cook County, IL. The primary questions it is designed to answer are:

1. Is the meditation app associated with improvements in behavioral health outcomes including cannabis use problems?
2. Do improvements in emotion regulation appear to mediate the effects of the meditation app on these behavioral health outcomes?
3. Will youth adequately adhere to the meditation app?

DETAILED DESCRIPTION:
This remote study will enroll 300 youth on probation in Cook County, IL, which encompasses Chicago and its surrounding suburbs. Youth will be individually randomized to use either the meditation app or an active control app matched for time/structure daily for 30 days. Health outcomes will be self-reported at baseline, 1 month, and 6 months, and in real time via 1-week "bursts" of ecological momentary assessment (EMA) at baseline and 1 month (i.e., approximately overlapping with the last week of app use). Objective adherence to both apps will be captured automatically via in-app analytics.

ELIGIBILITY:
Inclusion Criteria:

* 13-20 years old
* In probation programming (i.e., in legal programming but not detained) in Cook County
* Have access to an Apple/Android smartphone
* Understand and provide assent/consent
* Have parental consent (if under 18 years old)
* English-speaking, due to norming of instruments

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2029-08-30 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
Cannabis use problems | baseline, 1 month, 6 months
  The Cannabis Use Disorder Identification Test - Revised (CUDIT-R) includes 8 items, each rated on a 4-point scale; higher total scores indicate greater cannabis use problems
App adherence | 1 month
  App files played per objective in-app analytics data

SECONDARY OUTCOMES:
Sexual behaviors | baseline, 1 month, 6 months
  A modified AIDS Risk Behavior Assessment (ARBA) will be used to create a sexual behavior summary score; higher scores indicate more sexual risk behaviors
Negative mood regulation | baseline, 1 month, 6 months
  The Negative Mood Regulation (NMR) scale includes 14 items, each rated on a 5-point scale; higher total scores indicate greater beliefs one can regulate negative mood states
Anxiety | baseline, 1 month, 6 months
  The PROMIS Pediatric Item Bank GenPop v3.0 is a computer adaptive measure of anxiety; higher total scores indicate greater anxiety symptoms
Depression | baseline, 1 month, 6 months
  The PROMIS Pediatric Item Bank GenPop v3.0 is a computer adaptive measure of depression; higher total scores indicate greater depression symptoms
Self-efficacy | baseline, 1 month, 6 months
  The PROMIS Pediatric Item Bank GenPop v3.0 is a computer adaptive measure of self-efficacy; higher total scores indicate greater sense of self-efficacy
Alcohol use problems | baseline, 1 month, 6 months
  The Alcohol Trouble Scale (ATS) includes 10 items, each rated on a binary (yes/no) scale; higher scores indicate greater alcohol use problems
Real-time mood states | baseline, 1 month
  The International Positive Affect Negative Affect Schedule Short Form (I-PANAS-SF) includes 10 items, each rated on a 5-point scale; higher total scores indicate greater positive or negative moods, respectively at the time of ecological momentary assessment (EMA)
Real-time cannabis use | baseline, 1 month
  2 items indicating yes/no to cannabis use (1) now and (2) in the past 3 hours at the time of ecological momentary assessment (EMA)
Real-time alcohol use | baseline, 1 month
  2 items indicating yes/no to alcohol use (1) now and (2) in the past 3 hours at the time of ecological momentary assessment (EMA)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be placed in one or more electronic databases which could be used for other research studies.
Time Frame: Data sharing will generally coincide with publication of the study's main findings and is intended to take place within 1 year after acceptance of the primary manuscripts.
Access Criteria: To be determined